CLINICAL TRIAL: NCT00137046
Title: Efficacy and Safety of Exubera (Inhaled Insulin) Compared With Subcutaneous Human Insulin Therapy in Adult Subjects With Type 1 Diabetes Mellitus: A Long-Term, Outpatient, Open-Label, Parallel-Group Comparative Trial
Brief Title: Efficacy and Safety of Inhaled Insulin Compared With Subcutaneous Human Insulin Therapy in Adults With Type 1 Diabetes
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A2171022
Record Dates: First submitted 2005-08-26; First posted 2005-08-29 (Estimated); Results first posted 2010-01-26 (Estimated); Last update posted 2010-02-18 (Estimated); Status verified 2009-12

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Subcutaneous Insulin (Active Comparator)
  Interventions: Drug: Subcutaneous Insulin
- Inhaled Insulin (Experimental)
  Interventions: Drug: Inhaled Insulin

INTERVENTIONS:
Drug: Subcutaneous Insulin — Subcutaneous insulin with dose adjusted according to premeal blood glucose
  Arms: Subcutaneous Insulin
Drug: Inhaled Insulin — Inhaled insulin with dose adjusted according to premeal blood glucose
  Arms: Inhaled Insulin

SUMMARY:
This study is being done to find out the good and bad effects of a drug that is not approved for sale and the effects if any on measures of pulmonary function in adult males and females with type 1 diabetes mellitus. The drug is called EXUBERA (inhaled insulin).

This study included a 2-year comparative treatment period followed by a 6-month follow-up period during which inhaled insulin-treated subjects were switched back to subcutaneous short-acting insulin. After this follow-up period, all eligible subjects entered a comparative extension period that was to last for 5 years. When the comparative portion of the study was terminated, all subjects were requested to return for a final extension follow-up month 3 visit.

DETAILED DESCRIPTION:
Pfizer announced in October 2007 that it would stop marketing Exubera. Nektar, the company from which Pfizer licensed Exubera, announced on April 9, 2008 that it had stopped its search for a new marketing partner. Accordingly, there will be no commercial availability of Exubera. As a result, study A2171022 was terminated on June 9, 2008. Neither safety nor efficacy reasons were the cause of the study termination.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes mellitus

Exclusion Criteria:

* severe asthma or COPD
* smoking
* brittle diabetes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 582 (Actual)
Dates: Start 2002-05; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (60):
- United States (34):
  - Pfizer Investigational Site, Fullerton, California
  - Pfizer Investigational Site, Long Beach, California
  - Pfizer Investigational Site, Sacramento, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Santa Barbara, California
  - Pfizer Investigational Site, Santa Rosa, California
  - Pfizer Investigational Site, Tustin, California
  - Pfizer Investigational Site, Walnut Creek, California
  - Pfizer Investigational Site, Denver, Colorado
  - Pfizer Investigational Site, Longmont, Colorado
  - Pfizer Investigational Site, Hamden, Connecticut
  - Pfizer Investigational Site, Madison, Connecticut
  - Pfizer Investigational Site, Newark, Delaware
  - Pfizer Investigational Site, Coral Gables, Florida
  - Pfizer Investigational Site, Hollywood, Florida
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Tallahassee, Florida
  - Pfizer Investigational Site, West Palm Beach, Florida
  - Pfizer Investigational Site, Winter Park, Florida
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Wilmette, Illinois
  - Pfizer Investigational Site, Bethesda, Maryland
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Butte, Montana
  - Pfizer Investigational Site, New Hyde Park, New York
  - Pfizer Investigational Site, Durham, North Carolina
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Lansdale, Pennsylvania
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Burlington, Vermont
  - Pfizer Investigational Site, Richmond, Virginia
  - Pfizer Investigational Site, Renton, Washington
  - Pfizer Investigational Site, Milwaukee, Wisconsin
- Pfizer Investigational Site, Capital Federal, Buenos Aires, Argentina
- Brazil (5):
  - Pfizer Investigational Site, Belo Horizonte, Minas Gerais
  - Pfizer Investigational Site, Curitiba, Paraná
  - Pfizer Investigational Site, Porto Alegre, Rio Grande do Sul
  - Pfizer Investigational Site, Campinas, São Paulo
  - Pfizer Investigational Site, São Paulo, São Paulo
- Canada (17):
  - Pfizer Investigational Site, Calgary, Alberta
  - Pfizer Investigational Site, Edmonton, Alberta
  - Pfizer Investigational Site, Victoria, British Columbia
  - Pfizer Investigational Site, Winnepeg, Manitoba
  - Pfizer Investigational Site, Winnipeg, Manitoba
  - Pfizer Investigational Site, Halifax, Nova Scotia
  - Pfizer Investigational Site, Kingston, Ontario
  - Pfizer Investigational Site, London, Ontario
  - Pfizer Investigational Site, Mississauga, Ontario
  - Pfizer Investigational Site, Oakville, Ontario
  - Pfizer Investigational Site, Ottawa, Ontario
  - Pfizer Investigational Site, Thornhill, Ontario
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, Laval, Quebec
  - Pfizer Investigational Site, Montreal, Quebec
  - Pfizer Investigational Site, Sherbrooke, Quebec
  - Pfizer Investigational Site, Saskatoon, Saskatchewan
- Mexico (3):
  - Pfizer Investigational Site, Mexico City, COL LAS Americas
  - Pfizer Investigational Site, Mexico City, Mexico City
  - Pfizer Investigational Site, Monterrey, Nuevo León

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A2171022&StudyName=Efficacy%20and%20Safety%20of%20Inhaled%20Insulin%20Compared%20with%20Subcutaneous%20Human%20Insulin%20Therapy%20in%20Adults%20with%20Type%201%20Diabetes

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 64 centers took part in the study between 09 May 2002 and 08 December 2008.
Pre-assignment Details: At the screening visit and during the 4-week run-in phase all subjects received a subcutaneous insulin regimen consisting of 2 to 3 doses per day of regular insulin or short-acting insulin analog (lispro or aspart) plus 1 or 2 doses daily of intermediate-/long-acting insulin (NPH insulin or Ultralente), or insulin glargine once daily at bedtime.
Groups:
- Inhaled Insulin: Inhaled insulin (Exubera®) with dose adjusted according to premeal blood glucose plus basal insulin.
- Subcutaneous Insulin: Subcutaneous insulin with dose adjusted according to premeal blood glucose plus basal insulin.
Period: Overall Study
Arm/Group | Inhaled Insulin | Subcutaneous Insulin
Started | 291 (One subject was randomized to inhaled insulin but never received treatment.) | 291 (One subject was randomized to subcutaneous insulin but never received treatment.)
Received Study Treatment | 290 | 290
Completed | 192 (Completed subjects were those subjects who did not discontinue while on active drug.) | 198
Not Completed | 99 | 93
Not completed — Death | 2 | 1
Not completed — Adverse Event | 16 | 5
Not completed — Laboratory Abnormality | 2 | 0
Not completed — Lack of Efficacy | 13 | 1
Not completed — Lost to Follow-up | 8 | 24
Not completed — Other | 23 | 19
Not completed — Withdrawal by Subject | 33 | 42
Not completed — Adverse Event 4 Days after Last Dose | 1 | 0
Not completed — Withdrew prior to study treatment | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Inhaled Insulin | Subcutaneous Insulin | Total
Number analyzed (Participants) | 290 | 290 | 580
Age, Customized [Number; unit: years]
  18 to 25 | 48 | 53 | 101
  26 to 35 | 81 | 96 | 177
  36 to 45 | 94 | 71 | 165
  46 to 55 | 52 | 48 | 100
  56 to 65 | 15 | 22 | 37
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 121 | 129 | 250
  Male | 169 | 161 | 330

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Forced Expiratory Volume in One Second (FEV1)
Description: Change from Baseline: mean of (value of observed forced expiratory volume in the first second of forced exhalation [FEV1] in liters [L] at observation minus Baseline value).
Time Frame: Baseline through Extension Follow-up Month 3
Population: Full Analysis Set (FAS) FEV1: received at least 1 dose of study drug, had a Baseline FEV1, and at least 1 post-baseline FEV1. Due to study termination, originally planned inferential analysis for change from Month 3 through extension Month 60 was not done. Cross reference outcome measure: change from baseline in FEV1.
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Inhaled Insulin | Subcutaneous Insulin
Number analyzed (Participants) | 283 | 281
liters
  Baseline (n=283, 281) | 3.51 (0.76) | 3.47 (0.78)
  Month 3 (n=277, 263) | -0.04 (0.12) | -0.01 (0.12)
  Month 6 (n=262, 273) | -0.05 (0.14) | -0.03 (0.13)
  Month 9 (n=251, 264) | -0.06 (0.14) | -0.04 (0.13)
  Month 12 (n=242, 259) | -0.08 (0.14) | -004 (0.13)
  Month 15 (n=236, 250) | -0.09 (0.16) | -0.05 (0.15)
  Month 18 (n=227, 232) | -0.09 (0.15) | -0.06 (0.15)
  Month 21 (n=218, 224) | -0.11 (0.16) | -0.06 (0.15)
  Month 24 (n=211, 219) | -0.12 (0.17) | -0.08 (0.16)
  Follow-up Month 1 (n=242, 209) | -0.11 (0.17) | -0.09 (0.16)
  Follow-up Month 3 (n=249, 225) | -0.10 (0.16) | -0.09 (0.15)
  Follow-up Month 6 (n=240, 218) | -0.10 (0.17) | -0.09 (0.16)
  Extension Month 1 (n=166, 175) | -0.14 (0.20) | -0.10 (0.17)
  Extension Month 3 (n=161, 175) | -0.14 (0.18) | -0.10 (0.18)
  Extension Month 6 (n=158, 170) | -0.15 (0.19) | -0.11 (0.17)
  Extension Month 9 (n=151, 164) | -0.16 (0.18) | -0.12 (0.19)
  Extension Month 12 (n=152,161) | -0.17 (0.19) | -0.11 (0.16)
  Extension Month 15 (n=153,162) | -0.16 (0.19) | -0.12 (0.17)
  Extension Month 18 (n=148,160) | -0.18 (0.20) | -0.14 (0.19)
  Extension Month 21 (n=144,158) | -0.17 (0.19) | -0.15 (0.20)
  Extension Month 24 (n=141,153) | -0.18 (0.20) | -0.14 (0.20)
  Extension Month 27 (n=136,146) | -0.19 (0.20) | -0.13 (0.19)
  Extension Month 30 (n=136,147) | -0.20 (0.20) | -0.16 (0.19)
  Extension Month 33 (n=127,139) | -0.20 (0.21) | -0.17 (0.19)
  Extension Month 36 (n=105,126) | -0.23 (0.22) | -0.16 (0.18)
  Extension Month 39 (n=52, 64) | -0.21 (0.23) | -0.17 (0.21)
  Extension Month 39 (LOCF) (n=177, 187) | -0.22 (0.21) | -0.15 (0.19)
  Extension Follow Up Month 3 (n=115,102) | -0.20 (0.20) | -0.17 (0.18)
Statistical Analysis 1: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Month 3; Treatment difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted (Primary Analysis Model) includes terms of Treatment, Baseline Pulmonary Function Test (PFT), Center, Age, Sex, and Height; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.024, 90% CI [-0.041 to -0.007], Standard Error of Mean 0.010
Statistical Analysis 2: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Month 6; Treatment difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted (Primary Analysis Model) includes terms of Treatment, Baseline Pulmonary Function Test (PFT), Center, Age, Sex, and Height; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.022, 90% CI [-0.040 to -0.003], Standard Error of Mean 0.011
Statistical Analysis 3: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Month 9; Treatment difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted (Primary Analysis Model) includes terms of Treatment, Baseline Pulmonary Function Test (PFT), Center, Age, Sex, and Height; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.019, 90% CI [-0.038 to 0.001], Standard Error of Mean 0.012
Statistical Analysis 4: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Month 12; Treatment difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted (Primary Analysis Model) includes terms of Treatment, Baseline Pulmonary Function Test (PFT), Center, Age, Sex, and Height; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.038, 90% CI [-0.058 to -0.019], Standard Error of Mean 0.012
Statistical Analysis 5: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Month 15; Treatment difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted (Primary Analysis Model) includes terms of Treatment, Baseline Pulmonary Function Test (PFT), Center, Age, Sex, and Height; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.042, 90% CI [-0.065 to -0.020], Standard Error of Mean 0.014
Statistical Analysis 6: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Month 18; Treatment difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted (Primary Analysis Model) includes terms of Treatment, Baseline Pulmonary Function Test (PFT), Center, Age, Sex, and Height; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.020, 90% CI [-0.043 to 0.002], Standard Error of Mean 0.014
Statistical Analysis 7: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Month 21; Treatment difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted (Primary Analysis Model) includes terms of Treatment, Baseline Pulmonary Function Test (PFT), Center, Age, Sex, and Height; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.043, 90% CI [-0.066 to -0.020], Standard Error of Mean 0.014
Statistical Analysis 8: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Month 24; Treatment difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted (Primary Analysis Model) includes terms of Treatment, Baseline Pulmonary Function Test (PFT), Center, Age, Sex, and Height; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.033, 90% CI [-0.058 to -0.009], Standard Error of Mean 0.015
Statistical Analysis 9: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Follow-up Month 1; Treatment difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted (Primary Analysis Model) includes terms of Treatment, Baseline Pulmonary Function Test (PFT), Center, Age, Sex, and Height; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.015, 90% CI [-0.039 to 0.009], Standard Error of Mean 0.015
Statistical Analysis 10: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Follow-up Month 3; Treatment difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted (Primary Analysis Model) includes terms of Treatment, Baseline Pulmonary Function Test (PFT), Center, Age, Sex, and Height; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.005, 90% CI [-0.027 to 0.017], Standard Error of Mean 0.014
Statistical Analysis 11: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Follow-up Month 6; Treatment difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted (Primary Analysis Model) includes terms of Treatment, Baseline Pulmonary Function Test (PFT), Center, Age, Sex, and Height; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.013, 90% CI [-0.037 to 0.012], Standard Error of Mean 0.015
Statistical Analysis 12: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Extension Month 1; Treatment difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted (Primary Analysis Model) includes terms of Treatment, Baseline Pulmonary Function Test (PFT), Center, Age, Sex, and Height; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.045, 90% CI [-0.076 to -0.014], Standard Error of Mean 0.019
Statistical Analysis 13: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Extension Month 3; Treatment difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted (Primary Analysis Model) includes terms of Treatment, Baseline Pulmonary Function Test (PFT), Center, Age, Sex, and Height; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.045, 90% CI [-0.076 to -0.013], Standard Error of Mean 0.019
Statistical Analysis 14: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Extension Month 6; Treatment difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted (Primary Analysis Model) includes terms of Treatment, Baseline Pulmonary Function Test (PFT), Center, Age, Sex, and Height; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.040, 90% CI [-0.071 to -0.008], Standard Error of Mean 0.019
Statistical Analysis 15: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Extension Month 9; Treatment difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted (Primary Analysis Model) includes terms of Treatment, Baseline Pulmonary Function Test (PFT), Center, Age, Sex, and Height; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.041, 90% CI [-0.074 to -0.008], Standard Error of Mean 0.020
Statistical Analysis 16: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Extension Month 12; Treatment difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted (Primary Analysis Model) includes terms of Treatment, Baseline Pulmonary Function Test (PFT), Center, Age, Sex, and Height; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.056, 90% CI [-0.088 to -0.025], Standard Error of Mean 0.019
Statistical Analysis 17: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Extension Month 15; Treatment difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted (Primary Analysis Model) includes terms of Treatment, Baseline Pulmonary Function Test (PFT), Center, Age, Sex, and Height; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.039, 90% CI [-0.071 to -0.007], Standard Error of Mean 0.019
Statistical Analysis 18: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Extension Month 18; Treatment difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted (Primary Analysis Model) includes terms of Treatment, Baseline Pulmonary Function Test (PFT), Center, Age, Sex, and Height; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.044, 90% CI [-0.079 to -0.010], Standard Error of Mean 0.021
Statistical Analysis 19: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Extension Month 21; Treatment difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted (Primary Analysis Model) includes terms of Treatment, Baseline Pulmonary Function Test (PFT), Center, Age, Sex, and Height; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.020, 90% CI [-0.055 to 0.016], Standard Error of Mean 0.022
Statistical Analysis 20: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Extension Month 24; Treatment difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted (Primary Analysis Model) includes terms of Treatment, Baseline Pulmonary Function Test (PFT), Center, Age, Sex, and Height; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.042, 90% CI [-0.079 to -0.004], Standard Error of Mean 0.022
Statistical Analysis 21: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Extension Month 27; Treatment difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted (Primary Analysis Model) includes terms of Treatment, Baseline Pulmonary Function Test (PFT), Center, Age, Sex, and Height; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.055, 90% CI [-0.091 to -0.019], Standard Error of Mean 0.022
Statistical Analysis 22: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Extension Month 30; Treatment difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted (Primary Analysis Model) includes terms of Treatment, Baseline Pulmonary Function Test (PFT), Center, Age, Sex, and Height; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.045, 90% CI [-0.081 to -0.010], Standard Error of Mean 0.022
Statistical Analysis 23: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Extension Month 33; Treatment difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted (Primary Analysis Model) includes terms of Treatment, Baseline Pulmonary Function Test (PFT), Center, Age, Sex, and Height; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.036, 90% CI [-0.073 to 0.002], Standard Error of Mean 0.023
Statistical Analysis 24: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Extension Month 36; Treatment difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted (Primary Analysis Model) includes terms of Treatment, Baseline Pulmonary Function Test (PFT), Center, Age, Sex, and Height; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.079, 90% CI [-0.121 to -0.038], Standard Error of Mean 0.025
Statistical Analysis 25: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Extension Month 39; Treatment difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted (Primary Analysis Model) includes terms of Treatment, Baseline Pulmonary Function Test (PFT), Center, Age, Sex, and Height; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.061, 90% CI [-0.124 to 0.003], Standard Error of Mean 0.038
Statistical Analysis 26: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Extension Month 39 (LOCF); Treatment difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted (Primary Analysis Model) includes terms of Treatment, Baseline Pulmonary Function Test (PFT), Center, Age, Sex, and Height; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.066, 90% CI [-0.098 to -0.033], Standard Error of Mean 0.020
Statistical Analysis 27: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Extension Follow Up Month 3; Treatment difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted (Primary Analysis Model) includes terms of Treatment, Baseline Pulmonary Function Test (PFT), Center, Age, Sex, and Height; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.044, 90% CI [-0.085 to -0.004], Standard Error of Mean 0.024

2. Primary Outcome: Summary of ≥ 15% Decliners in Forced Expiratory Volume in One Second (FEV1)
Description: Number of subjects with a post-baseline Forced Expiratory Volume in One Second (FEV1) decrease of ≥ 15 % [(baseline observed value minus visit observed value)/(baseline observed value) * 100]; in the absence of an obvious intercurrent illness, a repeat FEV1 was performed.
Time Frame: Month 3 through Extension Follow-up 3
Population: FAS FEV1; (n) = number of subjects with analyzable data at observation for inhaled insulin and SC insulin, respectively.
Measure: Number; unit: participants
Arm/Group | Inhaled Insulin | Subcutaneous Insulin
Number analyzed (Participants) | 283 | 281
participants
  Month 3 (n=277, 263) | 0 | 0
  Month 6 (n=262, 273) | 0 | 0
  Month 9 (n=251, 264) | 0 | 1
  Month 12 (n=242, 259) | 1 | 0
  Month 15 (n=236, 250) | 3 | 1
  Month 18 (n=227, 232) | 0 | 3
  Month 21 (n=218, 224) | 2 | 3
  Month 24 (n=211, 219) | 3 | 2
  Follow-up Month 1 (n=242, 209) | 2 | 2
  Follow-up Month 3 (n=249, 225) | 3 | 3
  Follow-up Month 6 (n=240, 218) | 5 | 1
  Extension Month 1 (n=166, 175) | 2 | 2
  Extension Month 3 (n=161, 175) | 4 | 2
  Extension Month 6 (n=158, 170) | 2 | 2
  Extension Month 9 (n=151, 164) | 3 | 2
  Extension Month 12 (n=152, 161) | 2 | 0
  Extension Month 15 (n=153, 162) | 1 | 0
  Extension Month 18 (n=148, 160) | 4 | 3
  Extension Month 21 (n=144, 158) | 4 | 5
  Extension Month 24 (n=141, 153) | 3 | 5
  Extension Month 27 (n=136, 146) | 6 | 4
  Extension Month 30 (n=136, 147) | 6 | 2
  Extension Month 33 (n=127, 139) | 4 | 3
  Extension Month 36 (n=105, 126) | 7 | 3
  Extension Month 39 (n=52, 64) | 2 | 1
  Extension Follow Up Month 3 (n=115, 102) | 5 | 1

3. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1c)
Description: Change from Baseline: mean of (value of Glycosylated Hemoglobin [HbA1c] at observation minus Baseline value).
Time Frame: Baseline through Extension Follow-up Month 3
Population: FAS HbA1c: received at least 1 dose of study treatment, had baseline HbA1c and at least 1 post-baseline HbA1c; (n) = number of subjects with analyzable data at observation for inhaled insulin and SC insulin, respectively.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Inhaled Insulin | Subcutaneous Insulin
Number analyzed (Participants) | 288 | 286
percent
  Baseline (n=288, 286) | 7.41 (1.06) | 7.46 (1.06)
  Week 6 (n=269, 256) | -0.40 (0.61) | -0.43 (0.61)
  Month 3 (n=276, 280) | -0.36 (0.78) | -0.41 (0.73)
  Month 6 (n=263, 274) | -0.21 (0.80) | -0.36 (0.81)
  Month 9 (n=253, 266) | -0.10 (0.84) | -0.23 (0.81)
  Month 12 (n=240, 262) | -0.04 (0.87) | -0.32 (0.82)
  Month 15 (n=236, 253) | -0.12 (0.85) | -0.29 (0.90)
  Month 18 (n=231, 237) | -0.11 (0.88) | -0.30 (0.89)
  Month 21 (n=223, 231) | -0.05 (0.92) | -0.25 (0.92)
  Month 24 (n=214, 225) | 0.05 (0.91) | -0.27 (0.83)
  Follow-up Month 3 (n=205, 195) | -0.13 (0.87) | -0.22 (0.83)
  Follow-up Month 6 (n=219, 221) | -0.10 (0.87) | -0.14 (0.87)
  Extension Month 1 (n=171, 177) | -0.09 (0.90) | -0.23 (0.85)
  Extension Month 3 (n=170, 177) | 0.12 (0.95) | -0.17 (0.91)
  Extension Month 6 (n=166, 178) | 0.21 (0.99) | -0.19 (0.86)
  Extension Month 9 (n=159, 171) | 0.26 (1.00) | -0.06 (0.94)
  Extension Month 12 (n=158, 169) | 0.39 (0.98) | 0.08 (0.87)
  Extension Month 15 (n=156, 167) | 0.40 (1.05) | 0.17 (0.85)
  Extension Month 18 (n=153, 166) | 0.32 (0.94) | 0.05 (0.86)
  Extension Month 21 (n=154, 161) | 0.27 (0.99) | 0.00 (0.88)
  Extension Month 24 (n=149, 154) | 0.29 (0.89) | 0.06 (0.91)
  Extension Month 27 (n=141, 151) | 0.33 (0.97) | 0.10 (0.92)
  Extension Month 30 (n=140, 150) | 0.33 (0.91) | -0.01 (0.89)
  Extension Month 33 (n=131, 143) | 0.40 (0.94) | -0.08 (0.92)
  Extension Month 36 (n=108, 132) | 0.30 (0.99) | -0.03 (0.99)
  Extension Month 39 (n=55, 66) | 0.30 (0.94) | -0.09 (1.00)
  Extension Follow-Up Month 3 (n=120, 107) | 0.14 (1.00) | 0.12 (1.00)
Statistical Analysis 1: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Month 3; Treatment Difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted model includes terms of Treatment, Baseline HbA1c, and Center; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.031, 90% CI [-0.060 to 0.122], Standard Error of Mean 0.055
Statistical Analysis 2: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Month 6; Treatment Difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted model includes terms of Treatment, Baseline HbA1c, and Center; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.136, 90% CI [0.033 to 0.239], Standard Error of Mean 0.062
Statistical Analysis 3: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Month 9; Treatment Difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted model includes terms of Treatment, Baseline HbA1c, and Center; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.112, 90% CI [-0.000 to 0.224], Standard Error of Mean 0.068
Statistical Analysis 4: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Month 12; Treatment Difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted model includes terms of Treatment, Baseline HbA1c, and Center; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.257, 90% CI [0.141 to 0.374], Standard Error of Mean 0.071
Statistical Analysis 5: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Month 15; Treatment Difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted model includes terms of Treatment, Baseline HbA1c, and Center; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.156, 90% CI [0.040 to 0.273], Standard Error of Mean 0.071
Statistical Analysis 6: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Month 18; Treatment Difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted model includes terms of Treatment, Baseline HbA1c, and Center; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.182, 90% CI [0.065 to 0.300], Standard Error of Mean 0.072
Statistical Analysis 7: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Month 21; Treatment Difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted model includes terms of Treatment, Baseline HbA1c, and Center; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.190, 90% CI [0.060 to 0.319], Standard Error of Mean 0.078
Statistical Analysis 8: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Month 24; Treatment Difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted model includes terms of Treatment, Baseline HbA1c, and Center; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.316, 90% CI [0.190 to 0.443], Standard Error of Mean 0.077
Statistical Analysis 9: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Follow-up Month 3; Treatment Difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted model includes terms of Treatment, Baseline HbA1c, and Center; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.093, 90% CI [-0.037 to 0.224], Standard Error of Mean 0.079
Statistical Analysis 10: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Follow-up Month 6; Treatment Difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted model includes terms of Treatment, Baseline HbA1c, and Center; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.021, 90% CI [-0.103 to 0.145], Standard Error of Mean 0.075
Statistical Analysis 11: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Extension Month 1; Treatment Difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted model includes terms of Treatment, Baseline HbA1c, and Center; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.112, 90% CI [-0.023 to 0.248], Standard Error of Mean 0.082
Statistical Analysis 12: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Extension Month 3; Treatment Difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted model includes terms of Treatment, Baseline HbA1c, and Center; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.273, 90% CI [0.126 to 0.419], Standard Error of Mean 0.089
Statistical Analysis 13: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Extension Month 6; Treatment Difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted model includes terms of Treatment, Baseline HbA1c, and Center; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.363, 90% CI [0.219 to 0.507], Standard Error of Mean 0.087
Statistical Analysis 14: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Extension Month 9; Treatment Difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted model includes terms of Treatment, Baseline HbA1c, and Center; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.278, 90% CI [0.128 to 0.428], Standard Error of Mean 0.091
Statistical Analysis 15: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Extension Month 12; Treatment Difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted model includes terms of Treatment, Baseline HbA1c, and Center; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.293, 90% CI [0.144 to 0.442], Standard Error of Mean 0.091
Statistical Analysis 16: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Extension Month 15; Treatment Difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted model includes terms of Treatment, Baseline HbA1c, and Center; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.213, 90% CI [0.058 to 0.369], Standard Error of Mean 0.094
Statistical Analysis 17: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Extension Month 18; Treatment Difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted model includes terms of Treatment, Baseline HbA1c, and Center; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.243, 90% CI [0.101 to 0.386], Standard Error of Mean 0.086
Statistical Analysis 18: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Extension Month 21; Treatment Difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted model includes terms of Treatment, Baseline HbA1c, and Center; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.227, 90% CI [0.079 to 0.376], Standard Error of Mean 0.090
Statistical Analysis 19: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Extension Month 24; Treatment Difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted model includes terms of Treatment, Baseline HbA1c, and Center; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.225, 90% CI [0.079 to 0.372], Standard Error of Mean 0.089
Statistical Analysis 20: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Extension Month 27; Treatment Difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted model includes terms of Treatment, Baseline HbA1c, and Center; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.211, 90% CI [0.055 to 0.368], Standard Error of Mean 0.095
Statistical Analysis 21: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Extension Month 30; Treatment Difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted model includes terms of Treatment, Baseline HbA1c, and Center; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.331, 90% CI [0.180 to 0.483], Standard Error of Mean 0.092
Statistical Analysis 22: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Extension Month 33; Treatment Difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted model includes terms of Treatment, Baseline HbA1c, and Center; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.462, 90% CI [0.302 to 0.622], Standard Error of Mean 0.097
Statistical Analysis 23: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Extension Month 36; Treatment Difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted model includes terms of Treatment, Baseline HbA1c, and Center; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.410, 90% CI [0.221 to 0.600], Standard Error of Mean 0.115
Statistical Analysis 24: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Extension Month 39; Treatment Difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted model includes terms of Treatment, Baseline HbA1c, and Center; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.451, 90% CI [0.183 to 0.718], Standard Error of Mean 0.161
Statistical Analysis 25: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Extension Follow Up Month 3; Treatment Difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted model includes terms of Treatment, Baseline HbA1c, and Center; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.032, 90% CI [-0.174 to 0.237], Standard Error of Mean 0.124

4. Secondary Outcome: Hypoglycemic Event Rates
Description: A Hypoglycemic event was identified by characteristic symptoms of hypoglycemia with no blood glucose check with prompt resolution with food intake, subcutaneous glucagon, or intravenouus glucose; characteristic symptoms with blood glucose of 59 milligrams per deciliter (mg/dL) (3.2 mmol/L) or less with blood glucose check; or any glucose measurement of 49 mg/dL (2.7 mmol/L) or less, with or without symptoms. Subject months = elapsed number of months a subject was in the study in each time interval. Crude event rate = total events divided by subject month of treatment.
Time Frame: Month 1 through Extension Month 39
Population: FAS HbA1c; (n) = number of subjects with analyzable data at observation for inhaled insulin and SC insulin, respectively.
Measure: Number; unit: total events/subject months
Arm/Group | Inhaled Insulin | Subcutaneous Insulin
Number analyzed (Participants) | 288 | 286
total events/subject months
  Month 1 (n=288, 286) | 7.6 | 6.3
  Month 2 (n=282, 286) | 5.9 | 5.5
  Month 3 (n=279, 285) | 5.8 | 5.3
  Month 4 (n=273, 282) | 4.8 | 4.6
  Month 5 (n=266, 280) | 4.7 | 4.4
  Month 6 (n=263, 277) | 4.5 | 4.2
  Month 7 (n=259, 275) | 4.5 | 4.3
  Month 8 (n=257, 273) | 4.2 | 3.8
  Month 9 (n=254, 272) | 3.8 | 3.7
  Month 10 (n=249, 270) | 4.2 | 3.9
  Month 11 (n=245, 269) | 3.9 | 3.4
  Month 12 (n=243, 267) | 3.8 | 3.8
  Month 13 (n=239, 265) | 3.6 | 3.5
  Month 14 (n=237, 260) | 3.6 | 3.6
  Month 15 (n=236, 258) | 3.2 | 3.3
  Month 16 (n=236, 256) | 3.4 | 3.5
  Month 17 (n=235, 252) | 3.0 | 3.1
  Month 18 (n=233, 250) | 3.0 | 3.1
  Month 19 (n=232, 250) | 3.2 | 3.0
  Month 20 (n=227, 245) | 3.0 | 3.2
  Month 21 (n=226, 244) | 3.0 | 3.0
  Month 22 (n=226, 243) | 2.8 | 3.1
  Month 23 (n=224, 238) | 2.5 | 2.9
  Month 24 (n=222, 229) | 2.6 | 2.5
  Extension Month 1 (n=177, 187) | 3.5 | 2.9
  Extension Month 2 (n=177, 187) | 3.6 | 2.7
  Extension Month 3 (n=172, 185) | 4.1 | 2.9
  Extension Month 4 (n=169, 182) | 3.2 | 2.6
  Extension Month 5 (n=169, 182) | 3.2 | 2.8
  Extension Month 6 (n=168, 182) | 2.8 | 2.5
  Extension Month 7 (n=167, 181) | 3.1 | 2.5
  Extension Month 8 (n=167, 178) | 2.6 | 2.8
  Extension Month 9 (n=165, 177) | 2.1 | 2.6
  Extension Month 10 (n=165, 176) | 3.1 | 2.6
  Extension Month 11 (n=162, 175) | 3.2 | 2.2
  Extension Month 12 (n=160, 175) | 3.3 | 2.5
  Extension Month 13 (n=158, 174) | 2.8 | 2.6
  Extension Month 14 (n=156, 173) | 2.9 | 2.7
  Extension Month 15 (n=156, 173) | 3.0 | 2.3
  Extension Month 16 (n=156, 172) | 3.4 | 2.4
  Extension Month 17 (n=156, 172) | 3.0 | 2.3
  Extension Month 18 (n=156, 172) | 3.0 | 2.2
  Extension Month 19 (n=155, 172) | 3.2 | 2.6
  Extension Month 20 (n=155, 170) | 2.9 | 2.1
  Extension Month 21 (n=155, 169) | 2.8 | 2.3
  Extension Month 22 (n=155, 165) | 2.8 | 2.2
  Extension Month 23 (n=152, 164) | 3.3 | 2.3
  Extension Month 24 (n=152, 163) | 2.9 | 2.1
  Extension Month 25 (n=150, 162) | 3.2 | 2.1
  Extension Month 26 (n=149, 160) | 2.7 | 2.1
  Extension Month 27 (n=147, 159) | 2.7 | 1.9
  Extension Month 28 (n=146, 158) | 2.7 | 2.3
  Extension Month 29 (n=145, 155) | 2.7 | 2.0
  Extension Month 30 (n=143, 153) | 2.5 | 1.9
  Extension Month 31 (n=141, 153) | 2.6 | 2.2
  Extension Month 32 (n=138, 152) | 2.8 | 2.1
  Extension Month 33 (n=136, 150) | 2.3 | 2.1
  Extension Month 34 (n=131, 148) | 2.0 | 2.1
  Extension Month 35 (n=122, 147) | 1.8 | 2.1
  Extension Month 36 (n=113, 138) | 1.9 | 2.4
  Extension Month 37 (n=88, 104) | 1.5 | 2.0
  Extension Month 38 (n=66, 73) | 1.8 | 1.7
  Extension Month 39 (n=53, 64) | 1.7 | 1.4
  Overall Comparative (n=288, 286) | 4.1 | 3.9
  Overall Extension (n=177, 187) | 2.8 | 2.4

5. Secondary Outcome: Severe Hypoglycemic Event Rates
Description: Severe hypoglycemic event = all 3 of the following criteria were met: subject unable to treat self, exhbited at least 1 neurological symptom (memory loss, confusion, uncontrollable behavior, irrational behavior, unusual difficulty in awakening, suspected seizure, loss of consciousness); and blood glucose measurement was ≤49 mg/dL, or not measured but clinical manifestations reversed by oral carbohydrates, subcutaneous glucagon, or i.v. glucose. Subject months = elapsed number of months subject was in study in each time interval. Crude event rate = total events divided by subject months * 100.
Time Frame: Month 1 through Extension Month 39
Population: as for outcome 4
Measure: Number; unit: events / subject months * 100
Arm/Group | Inhaled Insulin | Subcutaneous Insulin
Number analyzed (Participants) | 288 | 286
events / subject months * 100
  Month 1 (n=288, 286) | 10.2 | 9.1
  Month 2 (n=282, 286) | 7.9 | 7.4
  Month 3 (n=279, 285) | 6.5 | 6.0
  Month 4 (n=273, 282) | 3.4 | 4.3
  Month 5 (n=266, 280) | 0.0 | 4.3
  Month 6 (n=263, 277) | 3.8 | 6.5
  Month 7 (n=259, 275) | 2.3 | 4.0
  Month 8 (n=257, 273) | 2.0 | 4.0
  Month 9 (n=254, 272) | 4.0 | 5.2
  Month 10 (n=249, 270) | 0.8 | 3.3
  Month 11 (n=245, 269) | 2.1 | 3.0
  Month 12 (n=243, 267) | 2.5 | 3.8
  Month 13 (n=239, 265) | 1.3 | 2.7
  Month 14 (n=237, 260) | 1.3 | 3.5
  Month 15 (n=236, 258) | 1.7 | 3.1
  Month 16 (n=236, 256) | 2.6 | 2.0
  Month 17 (n=235, 252) | 3.9 | 1.6
  Month 18 (n=233, 250) | 2.6 | 5.6
  Month 19 (n=232, 250) | 0.4 | 2.4
  Month 20 (n=227, 245) | 0.4 | 4.9
  Month 21 (n=226, 244) | 1.8 | 2.9
  Month 22 (n=226, 243) | 0.9 | 2.1
  Month 23 (n=224, 238) | 0.9 | 2.6
  Month 24 (n=222, 239) | 0.8 | 2.6
  Extension Month 1 (n=177, 187) | 3.9 | 1.2
  Extension Month 2 (n=177, 187) | 4.0 | 7.0
  Extension Month 3 (n=172, 185) | 4.0 | 2.4
  Extension Month 4 (n=169, 182) | 1.4 | 1.2
  Extension Month 5 (n=169, 182) | 2.7 | 4.2
  Extension Month 6 (n=168, 182) | 0.0 | 3.0
  Extension Month 7 (n=167, 181) | 0.7 | 2.4
  Extension Month 8 (n=167, 178) | 0.0 | 2.4
  Extension Month 9 (n=165, 177) | 2.1 | 4.9
  Extension Month 10 (n=165, 176) | 0.0 | 3.0
  Extension Month 11 (n=162, 175) | 2.8 | 1.2
  Extension Month 12 (n=160, 175) | 1.4 | 4.3
  Extension Month 13 (n=158, 174) | 0.7 | 1.8
  Extension Month 14 (n=156, 173) | 1.4 | 3.1
  Extension Month 15 (n=156, 173) | 1.4 | 11.1
  Extension Month 16 (n=156, 172) | 0.7 | 13.7
  Extension Month 17 (n=156, 172) | 0.7 | 5.6
  Extension Month 18 (n=156, 172) | 0.0 | 7.5
  Extension Month 19 (n=155, 172) | 1.4 | 6.9
  Extension Month 20 (n=155, 170) | 2.1 | 2.5
  Extension Month 21 (n=155, 169) | 1.4 | 3.8
  Extension Month 22 (n=155, 165) | 2.1 | 1.3
  Extension Month 23 (n=152, 164) | 1.4 | 3.2
  Extension Month 24 (n=152, 163) | 0.7 | 3.2
  Extension Month 25 (n=150, 162) | 1.5 | 0.0
  Extension Month 26 (n=149, 160) | 2.2 | 0.7
  Extension Month 27 (n=147, 159) | 0.7 | 0.0
  Extension Month 28 (n=146, 158) | 0.0 | 3.4
  Extension Month 29 (n=145, 155) | 0.0 | 0.7
  Extension Month 30 (n=143, 153) | 0.8 | 0.7
  Extension Month 31 (n=141, 153) | 3.1 | 0.0
  Extension Month 32 (n=138, 152) | 0.0 | 1.4
  Extension Month 33 (n=136, 150) | 2.4 | 1.4
  Extension Month 34 (n=131, 148) | 0.8 | 1.4
  Extension Month 35 (n=122, 147) | 0.0 | 5.9
  Extension Month 36 (n=113, 138) | 1.0 | 0.9
  Extension Month 37 (n=88, 104) | 0.0 | 3.8
  Extension Month 38 (n=66, 73) | 0.0 | 0.0
  Extension Month 39 (n=53, 64) | 0.8 | 1.7
  Overall Comparative (n=288, 286) | 2.8 | 4.1
  Overall Extension (n=177, 187) | 1.4 | 3.3

6. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose
Description: Change from Baseline: mean of (value of fasting plasma glucose [milligrams per deciliter (mg/dL)] at observation minus Baseline value).
Time Frame: Baseline through Extension Follow-up Month 3
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Inhaled Insulin | Subcutaneous Insulin
Number analyzed (Participants) | 286 | 286
mg/dL
  Baseline (n=286, 286) | 171.24 (63.20) | 170.06 (55.20)
  Week 6 (n=263, 250) | -26.04 (84.79) | -14.02 (80.13)
  Month 3 (n=267, 276) | -21.84 (85.26) | -6.15 (79.08)
  Month 6 (n=258, 271) | -31.48 (81.62) | -6.29 (83.81)
  Month 9 (n=243, 262) | -25.34 (86.24) | 1.28 (96.32)
  Month 12 (n=232, 256) | -24.25 (87.53) | -4.95 (85.96)
  Month 15 (n=230, 251) | -34.75 (83.72) | 5.96 (89.39)
  Month 18 (n=226, 236) | -24.13 (86.44) | -8.13 (88.83)
  Month 21 (n=216, 230) | -26.77 (88.96) | -11.62 (82.98)
  Month 24 (n=208, 222) | -18.36 (92.92) | 1.25 (84.87)
  Follow-up Month 3 (n=2, 2) | -43.50 (85.09) | 46.67 (24.04)
  Follow-up Month 6 (n=159, 164) | 3.45 (80.26) | 1.46 (85.49)
  Extension Month 1 (n=164, 171) | -25.52 (90.15) | -2.72 (91.27)
  Extension Month 3 (n=167, 172) | -25.02 (87.75) | 0.43 (84.55)
  Extension Month 6 (n=164, 177) | -13.47 (80.85) | -12.56 (86.93)
  Extension Month 9 (n=152, 170) | -16.19 (94.12) | -4.46 (88.86)
  Extension Month 12 (n=155, 167) | -22.53 (83.01) | -5.15 (81.38)
  Extension Month 15 (n=148, 163) | -26.11 (85.78) | -10.64 (86.00)
  Extension Month 18 (n=148, 163) | -12.42 (86.69) | -2.32 (84.41)
  Extension Month 21 (n=152, 157) | -24.75 (87.29) | 4.86 (89.31)
  Extension Month 24 (n=142, 148) | -20.46 (86.45) | -10.36 (93.08)
  Extension Month 27 (n=140, 148) | -14.91 (78.42) | -2.86 (91.97)
  Extension Month 30 (n=138, 147) | -17.16 (86.47) | -3.77 (86.15)
  Extension Month 33 (n=129, 141) | -22.77 (94.77) | -12.12 (88.26)
  Extension Month 36 (n=107, 132) | -20.00 (81.03) | -2.49 (86.06)
  Extension Month 39 (n=55, 64) | -38.47 (95.17) | -1.57 (78.47)
  Extension Follow-Up Month 3 (n=118, 105) | 1.97 (95.39) | 3.25 (84.53)
Statistical Analysis 1: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Month 3; Treatment Difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted model includes terms of Treatment, Baseline Fasting Plasma Glucose, and Center; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -14.81, 90% CI [-25.24 to -4.39], Standard Error of Mean 6.33
Statistical Analysis 2: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Month 6; Treatment Difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted model includes terms of Treatment, Baseline Fasting Plasma Glucose, and Center; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -24.83, 90% CI [-35.16 to -14.51], Standard Error of Mean 6.27
Statistical Analysis 3: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Month 9; Treatment Difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted model includes terms of Treatment, Baseline Fasting Plasma Glucose, and Center; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -26.16, 90% CI [-37.56 to -14.75], Standard Error of Mean 6.92
Statistical Analysis 4: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Month 12; Treatment Difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted model includes terms of Treatment, Baseline Fasting Plasma Glucose, and Center; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -19.46, 90% CI [-30.56 to -8.36], Standard Error of Mean 6.74
Statistical Analysis 5: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Month 15; Treatment Difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted model includes terms of Treatment, Baseline Fasting Plasma Glucose, and Center; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -39.97, 90% CI [-50.93 to -29.00], Standard Error of Mean 6.65
Statistical Analysis 6: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Month 18; Treatment Difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted model includes terms of Treatment, Baseline Fasting Plasma Glucose, and Center; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -16.08, 90% CI [-27.65 to -4.51], Standard Error of Mean 7.02
Statistical Analysis 7: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Month 21; Treatment Difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted model includes terms of Treatment, Baseline Fasting Plasma Glucose, and Center; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -13.54, 90% CI [-24.69 to -2.39], Standard Error of Mean 6.76
Statistical Analysis 8: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Month 24; Treatment Difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted model includes terms of Treatment, Baseline Fasting Plasma Glucose, and Center; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -18.86, 90% CI [-30.88 to -6.84], Standard Error of Mean 7.29
Statistical Analysis 9: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Follow-up Month 6; Treatment Difference: Inhaled Insulin - Subcutaneous Insulin.Adjusted model includes terms of Treatment, Baseline Fasting Plasma Glucose, and Center; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 3.56, 90% CI [-9.83 to 16.96], Standard Error of Mean 8.12
Statistical Analysis 10: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Extension Month 1; Treatment Difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted model includes terms of Treatment, Baseline Fasting Plasma Glucose, and Center; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -17.80, 90% CI [-31.32 to -4.27], Standard Error of Mean 8.20
Statistical Analysis 11: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Extension Month 3; Treatment Difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted model includes terms of Treatment, Baseline Fasting Plasma Glucose, and Center; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -20.71, 90% CI [-33.44 to -7.99], Standard Error of Mean 7.72
Statistical Analysis 12: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Extension Month 6; Treatment Difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted model includes terms of Treatment, Baseline Fasting Plasma Glucose, and Center; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 1.80, 90% CI [-11.06 to 14.66], Standard Error of Mean 7.80
Statistical Analysis 13: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Extension Month 9; Treatment Difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted model includes terms of Treatment, Baseline Fasting Plasma Glucose, and Center; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -8.72, 90% CI [-23.61 to 6.17], Standard Error of Mean 9.02
Statistical Analysis 14: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Extension Month 12; Treatment Difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted model includes terms of Treatment, Baseline Fasting Plasma Glucose, and Center; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -16.34, 90% CI [-29.28 to -3.40], Standard Error of Mean 7.84
Statistical Analysis 15: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Extension Month 15; Treatment Difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted model includes terms of Treatment, Baseline Fasting Plasma Glucose, and Center; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -12.99, 90% CI [-26.60 to 0.63], Standard Error of Mean 8.25
Statistical Analysis 16: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Extension Month 18; Treatment Difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted model includes terms of Treatment, Baseline Fasting Plasma Glucose, and Center; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -10.22, 90% CI [-24.39 to 3.94], Standard Error of Mean 8.58
Statistical Analysis 17: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Extension Month 21; Treatment Difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted model includes terms of Treatment, Baseline Fasting Plasma Glucose, and Center; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -28.64, 90% CI [-43.19 to -14.09], Standard Error of Mean 8.82
Statistical Analysis 18: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Extension Month 24; Treatment Difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted model includes terms of Treatment, Baseline Fasting Plasma Glucose, and Center; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -8.99, 90% CI [-23.69 to 5.71], Standard Error of Mean 8.91
Statistical Analysis 19: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Extension Month 27; Treatment Difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted model includes terms of Treatment, Baseline Fasting Plasma Glucose, and Center; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -9.52, 90% CI [-24.04 to 5.00], Standard Error of Mean 8.80
Statistical Analysis 20: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Extension Month 30; Treatment Difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted model includes terms of Treatment, Baseline Fasting Plasma Glucose, and Center; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -10.40, 90% CI [-24.71 to 3.92], Standard Error of Mean 8.67
Statistical Analysis 21: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Extension Month 33; Treatment Difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted model includes terms of Treatment, Baseline Fasting Plasma Glucose, and Center; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -6.17, 90% CI [-21.42 to 9.09], Standard Error of Mean 9.24
Statistical Analysis 22: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Extension Month 36; Treatment Difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted model includes terms of Treatment, Baseline Fasting Plasma Glucose, and Center; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -5.39, 90% CI [-20.98 to 10.21], Standard Error of Mean 9.44
Statistical Analysis 23: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Extension Month 39; Treatment Difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted model includes terms of Treatment, Baseline Fasting Plasma Glucose, and Center; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -15.58, 90% CI [-38.43 to 7.26], Standard Error of Mean 13.77
Statistical Analysis 24: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Extension Follow Up Month 3; Treatment Difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted model includes terms of Treatment, Baseline Fasting Plasma Glucose, and Center; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 2.84, 90% CI [-15.79 to 21.46], Standard Error of Mean 11.27

7. Secondary Outcome: Change From Baseline Body Weight
Description: Body weight: mean Baseline and change from Baseline in kilograms (kg). Change from baseline = mean body weight in kilograms (kg) at observation minus mean baseline body weight.
Time Frame: Baseline through Extension Follow-up Month 3
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Inhaled Insulin | Subcutaneous Insulin
Number analyzed (Participants) | 288 | 286
kilograms
  Baseline (n=288, 286) | 75.12 (13.57) | 73.72 (13.13)
  Week 4 (n=257, 247) | 0.30 (1.39) | 0.63 (3.01)
  Week 8 (n=263, 262) | 0.46 (1.88) | 0.67 (2.00)
  Month 3 (n=273, 269) | 0.13 (2.20) | 0.67 (2.35)
  Week 18 (n=248, 260) | 0.15 (2.60) | 1.00 (2.64)
  Month 6 (n=259, 272) | 0.11 (2.89) | 1.25 (3.08)
  Month 9 (n=251, 266) | 0.05 (3.28) | 1.41 (3.35)
  Month 12 (n=242, 259) | 0.37 (3.46) | 1.55 (3.59)
  Month 15 (n=236, 250) | 0.44 (3.57) | 1.84 (3.90)
  Month 18 (n=227, 233) | 0.57 (3.99) | 2.26 (4.30)
  Month 21 (n=220, 224) | 1.07 (4.22) | 2.35 (4.51)
  Month 24 (n=211, 220) | 0.99 (4.58) | 2.23 (4.58)
  Follow-up Month 3 (n=248, 225) | 1.50 (4.24) | 2.31 (4.89)
  Follow-up Month 6 (n=239, 219) | 1.68 (4.28) | 2.17 (4.46)
  Extension Month 1 (n=166, 175) | 2.44 (6.98) | 2.50 (4.93)
  Extension Month 3 (n=161, 175) | 1.73 (4.69) | 3.08 (7.17)
  Extension Month 6 (n=158, 170) | 1.67 (4.93) | 3.05 (4.75)
  Extension Month 9 (n=153, 164) | 1.61 (4.73) | 3.17 (5.27)
  Extension Month 12 (n=152, 162) | 2.11 (4.95) | 3.08 (4.93)
  Extension Month 15 (n=153, 162) | 2.01 (5.06) | 3.16 (5.21)
  Extension Month 18 (n=149, 160) | 2.31 (5.50) | 3.30 (5.82)
  Extension Month 21 (n=144, 158) | 2.14 (5.63) | 3.72 (5.82)
  Extension Month 24 (n=141, 153) | 2.49 (5.98) | 4.23 (5.70)
  Extension Month 27 (n=136, 146) | 2.12 (5.87) | 3.96 (6.15)
  Extension Month 30 (n=136, 147) | 2.42 (6.25) | 4.80 (8.38)
  Extension Month 33 (n=127, 139) | 2.30 (5.96) | 5.28 (10.84)
  Extension Month 36 (n=105, 126) | 2.11 (6.24) | 3.87 (6.25)
  Extension Month 39 (n=52, 64) | 1.58 (7.90) | 4.83 (6.75)
  Extension Follow-Up Month 3 (n=116, 103) | 2.49 (5.98) | 4.09 (6.34)
Statistical Analysis 1: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Month 3; Treatment-Difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted model includes terms of Treatment, Baseline Body Weight, and Center; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.523, 90% CI [-0.846 to -0.199], Standard Error of Mean 0.196
Statistical Analysis 2: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Month 6; Treatment-Difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted model includes terms of Treatment, Baseline Body Weight, and Center; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -1.113, 90% CI [-1.541 to -0.685], Standard Error of Mean 0.260
Statistical Analysis 3: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Month 9; Treatment-Difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted model includes terms of Treatment, Baseline Body Weight, and Center; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -1.359, 90% CI [-1.836 to -0.882], Standard Error of Mean 0.290
Statistical Analysis 4: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Month 12; Treatment-Difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted model includes terms of Treatment, Baseline Body Weight, and Center; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -1.184, 90% CI [-1.702 to -0.666], Standard Error of Mean 0.314
Statistical Analysis 5: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Month 15; Treatment-Difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted model includes terms of Treatment, Baseline Body Weight, and Center; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -1.426, 90% CI [-1.984 to -0.869], Standard Error of Mean 0.338
Statistical Analysis 6: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Month 18; Treatment-Difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted model includes terms of Treatment, Baseline Body Weight, and Center; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -1.717, 90% CI [-2.350 to -1.084], Standard Error of Mean 0.384
Statistical Analysis 7: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Month 21; Treatment-Difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted model includes terms of Treatment, Baseline Body Weight, and Center; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -1.273, 90% CI [-1.950 to -0.596], Standard Error of Mean 0.411
Statistical Analysis 8: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Month 24; Treatment-Difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted model includes terms of Treatment, Baseline Body Weight, and Center; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -1.069, 90% CI [-1.792 to -0.346], Standard Error of Mean 0.439
Statistical Analysis 9: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Follow-up Month 3; Treatment-Difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted model includes terms of Treatment, Baseline Body Weight, and Center; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.785, 90% CI [-1.475 to -0.096], Standard Error of Mean 0.418
Statistical Analysis 10: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Follow-up Month 6; Treatment-Difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted model includes terms of Treatment, Baseline Body Weight, and Center; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.445, 90% CI [-1.114 to 0.224], Standard Error of Mean 0.406
Statistical Analysis 11: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Extension Month 1; Treatment-Difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted model includes terms of Treatment, Baseline Body Weight, and Center; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.054, 90% CI [-1.133 to 1.025], Standard Error of Mean 0.654
Statistical Analysis 12: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Extension Month 3; Treatment-Difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted model includes terms of Treatment, Baseline Body Weight, and Center; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -1.336, 90% CI [-2.438 to -0.235], Standard Error of Mean 0.668
Statistical Analysis 13: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Extension Month 6; Treatment-Difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted model includes terms of Treatment, Baseline Body Weight, and Center; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -1.462, 90% CI [-2.356 to -0.568], Standard Error of Mean 0.542
Statistical Analysis 14: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Extension Month 9; Treatment-Difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted model includes terms of Treatment, Baseline Body Weight, and Center; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -1.385, 90% CI [-2.316 to -0.454], Standard Error of Mean 0.564
Statistical Analysis 15: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Extension Month 12; Treatment-Difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted model includes terms of Treatment, Baseline Body Weight, and Center; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.955, 90% CI [-1.877 to -0.034], Standard Error of Mean 0.559
Statistical Analysis 16: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Extension Month 15; Treatment-Difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted model includes terms of Treatment, Baseline Body Weight, and Center; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -1.000, 90% CI [-1.970 to -0.030], Standard Error of Mean 0.588
Statistical Analysis 17: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Extension Month 18; Treatment-Difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted model includes terms of Treatment, Baseline Body Weight, and Center; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.960, 90% CI [-2.041 to 0.121], Standard Error of Mean 0.655
Statistical Analysis 18: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Extension Month 21; Treatment-Difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted model includes terms of Treatment, Baseline Body Weight, and Center; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -1.667, 90% CI [-2.770 to -0.565], Standard Error of Mean 0.668
Statistical Analysis 19: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Extension Month 24; Treatment-Difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted model includes terms of Treatment, Baseline Body Weight, and Center; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -1.872, 90% CI [-3.013 to -0.730], Standard Error of Mean 0.692
Statistical Analysis 20: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Extension Month 27; Treatment-Difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted model includes terms of Treatment, Baseline Body Weight, and Center; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -1.887, 90% CI [-3.084 to -0.690], Standard Error of Mean 0.725
Statistical Analysis 21: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Extension Month 30; Treatment-Difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted model includes terms of Treatment, Baseline Body Weight, and Center; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -2.794, 90% CI [-4.264 to -1.324], Standard Error of Mean 0.891
Statistical Analysis 22: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Extension Month 33; Treatment-Difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted model includes terms of Treatment, Baseline Body Weight, and Center; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -3.287, 90% CI [-5.088 to -1.485], Standard Error of Mean 1.091
Statistical Analysis 23: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Extension Month 36; Treatment-Difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted model includes terms of Treatment, Baseline Body Weight, and Center; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -1.486, 90% CI [-2.901 to -0.071], Standard Error of Mean 0.857
Statistical Analysis 24: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Extension Month 39; Treatment-Difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted model includes terms of Treatment, Baseline Body Weight, and Center; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -3.131, 90% CI [-5.382 to -0.880], Standard Error of Mean 1.356
Statistical Analysis 25: Comparison: Inhaled Insulin vs Subcutaneous Insulin; Extension Follow Up Month 3; Treatment-Difference: Inhaled Insulin - Subcutaneous Insulin. Adjusted model includes terms of Treatment, Baseline Body Weight, and Center; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -1.487, 90% CI [-2.918 to -0.055], Standard Error of Mean 0.866

8. Secondary Outcome: Total Daily Long-Acting Insulin Dose (Unadjusted for Body Weight)
Description: Total Daily Long-Acting Insulin Dose Unadjusted for Body Weight; long-acting insulin included NPH Insulin, Ultralente, and Insulin Glargine for both groups.
Time Frame: Month 3 through Extension Month 39
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units
Arm/Group | Inhaled Insulin | Subcutaneous Insulin
Number analyzed (Participants) | 288 | 286
units
  Month 3 (n=280, 285) | 30.52 (16.00) | 34.97 (17.38)
  Month 6 (n=271, 280) | 30.57 (16.48) | 35.37 (17.72)
  Month 9 (n=256, 269) | 30.69 (16.53) | 35.35 (18.06)
  Month 12 (n=243, 262) | 30.65 (17.29) | 35.42 (18.00)
  Month 15 (n=237, 255) | 30.99 (17.83) | 35.75 (17.86)
  Month 18 (n=234, 242) | 30.97 (17.86) | 36.35 (18.13)
  Month 21 (n=224, 233) | 31.30 (18.53) | 36.75 (17.76)
  Month 24 (n=218, 229) | 31.82 (19.36) | 36.21 (18.02)
  Extension Month 1 (n=171, 178) | 32.84 (18.90) | 35.67 (18.72)
  Extension Month 3 (n=170, 177) | 32.45 (18.91) | 35.10 (18.07)
  Extension Month 6 (n=166, 179) | 31.96 (18.36) | 34.75 (17.55)
  Extension Month 9 (n=160, 174) | 32.73 (19.24) | 35.22 (17.41)
  Extension Month 12 (n=159, 169) | 32.29 (19.12) | 33.82 (15.65)
  Extension Month 15 (n=156, 164) | 32.02 (18.61) | 35.52 (18.37)
  Extension Month 18 (n=152, 166) | 32.37 (18.62) | 34.88 (17.44)
  Extension Month 21 (n=154, 165) | 31.83 (19.05) | 35.14 (17.24)
  Extension Month 24 (n=150, 153) | 31.99 (19.59) | 35.61 (18.34)
  Extension Month 27 (n=142, 153) | 31.25 (19.01) | 35.58 (18.42)
  Extension Month 30 (n=141, 148) | 31.06 (19.73) | 35.34 (18.73)
  Extension Month 33 (n=133, 144) | 30.71 (19.06) | 34.83 (17.47)
  Extension Month 36 (n=113, 136) | 29.62 (19.06) | 33.58 (15.64)
  Extension Month 39 (n=57, 67) | 29.07 (16.59) | 33.63 (19.79)

9. Secondary Outcome: Total Daily Long-Acting Insulin Dose Adjusted for Body Weight
Description: Total daily dose of long-acting insulin adjusted for body weight (units per kilogram [kg]). Long-acting insulin included NPH Insulin, Ultralente, and Insulin Glargine for both groups.
Time Frame: Month 3 through Extension Month 39
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units/kg
Arm/Group | Inhaled Insulin | Subcutaneous Insulin
Number analyzed (Participants) | 288 | 286
units/kg
  Month 3 (n=280, 285) | 0.41 (0.22) | 0.48 (0.25)
  Month 6 (n=271, 280) | 0.41 (0.23) | 0.49 (0.25)
  Month9 (n=256, 269) | 0.41 (0.23) | 0.49 (0.26)
  Month 12 (n=243, 262) | 0.41 (0.24) | 0.49 (0.26)
  Month 15 (n=237, 255) | 0.42 (0.25) | 0.49 (0.25)
  Month 18 (n=234, 242) | 0.42 (0.25) | 0.50 (0.26)
  Month 21 (n=224, 233) | 0.42 (0.26) | 0.51 (0.26)
  Month 24 (n=218, 229) | 0.43 (0.27) | 0.50 (0.26)
  Extension Month 1 (n=171, 178) | 0.45 (0.25) | 0.49 (0.27)
  Extension Month 3 (n=170, 177) | 0.44 (0.25) | 0.49 (0.26)
  Extension Month 6 (n=166, 179) | 0.43 (0.24) | 0.48 (0.26)
  Extension Month 9 (n=160, 174) | 0.44 (0.25) | 0.49 (0.25)
  Extension Month 12 (n=159, 169) | 0.44 (0.24) | 0.47 (0.22)
  Extension Month 15 (n=156, 164) | 0.44 (0.25) | 0.49 (0.26)
  Extension Month 18 (n=152, 166) | 0.44 (0.25) | 0.48 (0.24)
  Extension Month 21 (n=154, 165) | 0.44 (0.25) | 0.48 (0.23)
  Extension Month 24 (n=150, 153) | 0.44 (0.26) | 0.49 (0.25)
  Extension Month 27 (n=142, 153) | 0.43 (0.24) | 0.49 (0.24)
  Extension Month 30 (n=141, 148) | 0.42 (0.26) | 0.49 (0.26)
  Extension Month 33 (n=133, 144) | 0.42 (0.25) | 0.48 (0.23)
  Extension Month 36 (n=113, 136) | 0.40 (0.25) | 0.46 (0.21)
  Extension Month 39 (n=57, 67) | 0.39 (0.23) | 0.45 (0.25)

10. Secondary Outcome: Total Daily Short-Acting Insulin Dose (Unadjusted for Body Weight)
Description: Total daily dose of short-acting insulin unadjusted for body weight. Short-acting insulin (mg) for the Inhaled Insulin group was Inhaled Insulin. Short-acting insulin (unit) for the Subcutaneous Insulin group included Insulin Lispro, Insulin Aspart, and Regular Insulin.
Time Frame: Month 3 through Extension Month 39
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mg, units
Groups:
- Inhaled Insulin (mg): Inhaled insulin (Exubera®) with dose adjusted according to premeal blood glucose plus basal insulin.
- Subcutaneous Insulin (Units): Subcutaneous insulin with dose adjusted according to premeal blood glucose plus basal insulin.
Arm/Group | Inhaled Insulin (mg) | Subcutaneous Insulin (Units)
Number analyzed (Participants) | 288 | 286
mg, units
  Month 3 (n=280, 285) | 10.45 (5.71) | 25.05 (14.73)
  Month 6 (n=271, 281) | 11.50 (6.73) | 25.14 (14.72)
  Month 9 (n=257, 271) | 11.97 (6.79) | 24.90 (14.54)
  Month 12 (n=243, 266) | 12.69 (6.96) | 25.32 (14.35)
  Month 15 (n=237, 255) | 13.12 (7.65) | 25.11 (14.83)
  Month 18 (n=234, 241) | 13.60 (8.04) | 25.20 (15.15)
  Month 21 (n=224, 235) | 14.42 (8.64) | 25.45 (15.41)
  Month 24 (n=219, 232) | 14.61 (9.14) | 25.23 (16.57)
  Extension Month 1 (n=170, 179) | 11.49 (6.35) | 25.84 (17.48)
  Extension Month 3 (n=170, 178) | 12.50 (6.88) | 25.94 (18.26)
  Extension Month 6 (n=166, 179) | 13.64 (9.07) | 25.39 (17.52)
  Extension Month 9 (n=160, 174) | 14.06 (9.33) | 26.19 (18.00)
  Extension Month 12 (n=159, 169) | 14.74 (10.07) | 25.49 (17.69)
  Extension Month 15 (n=156, 167) | 13.93 (8.38) | 25.80 (17.62)
  Extension Month 18 (n=153, 167) | 13.97 (8.58) | 26.04 (17.52)
  Extension Month 21 (n=154, 166) | 14.53 (8.80) | 25.95 (17.04)
  Extension Month 24 (n=150, 156) | 14.48 (8.71) | 27.26 (19.48)
  Extension Month 27 (n=142, 153) | 14.82 (8.70) | 26.63 (17.82)
  Extension Month 30 (n=141, 149) | 14.92 (8.93) | 27.22 (18.66)
  Extension Month 33 (n=133, 144) | 15.28 (9.72) | 26.71 (18.67)
  Extension Month 36 (n=113, 136) | 15.72 (8.32) | 27.04 (19.65)
  Extension Month 39 (n=57, 67) | 17.92 (12.04) | 29.75 (19.68)

11. Secondary Outcome: Total Daily Short-Acting Insulin Dose Adjusted for Body Weight
Description: Total Daily Short-Acting Insulin Dose adjusted for body weight (milligrams [mg] or units divided by kilograms [kg]). Short-acting insulin (mg) for the Inhaled Insulin group was Inhaled Insulin. Short-acting insulin (unit) for the Subcutaneous Insulin group included Insulin Lispro, Insulin Aspart, and Regular Insulin.
Time Frame: Month 3 through Extension Month 39
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mg/kg, units/kg
Groups:
- Inhaled Insulin (mg/kg): Inhaled insulin (Exubera®) with dose adjusted according to premeal blood glucose plus basal insulin.
- Subcutaneous Insulin (Units/kg): Subcutaneous insulin with dose adjusted according to premeal blood glucose plus basal insulin.
Arm/Group | Inhaled Insulin (mg/kg) | Subcutaneous Insulin (Units/kg)
Number analyzed (Participants) | 288 | 286
mg/kg, units/kg
  Month 3 (n=280, 285) | 0.14 (0.07) | 0.34 (0.19)
  Month 6 (n=271, 281) | 0.15 (0.08) | 0.34 (0.19)
  Month 9 (n=257, 271) | 0.16 (0.09) | 0.34 (0.18)
  Month 12 (n=243, 266) | 0.17 (0.09) | 0.34 (0.18)
  Month 15 (n=237, 255) | 0.17 (0.10) | 0.34 (0.19)
  Month 18 (n=234, 241) | 0.18 (0.10) | 0.34 (0.19)
  Month 21 (n=224, 235) | 0.19 (0.11) | 0.34 (0.20)
  Month 24 (n=219, 232) | 0.19 (0.12) | 0.34 (0.21)
  Extension Month 1 (n=170, 179) | 0.15 (0.08) | 0.35 (0.22)
  Extension Month 3 (n=170, 178) | 0.17 (0.08) | 0.35 (0.23)
  Extension Month 6 (n=166, 179) | 0.18 (0.10) | 0.34 (0.22)
  Extension Month 9 (n=160, 174) | 0.19 (0.11) | 0.35 (0.22)
  Extension Month 12 (n=159, 169) | 0.20 (0.13) | 0.34 (0.22)
  Extension Month 15 (n=156, 167) | 0.19 (0.10) | 0.35 (0.22)
  Extension Month 18 (n=153, 167) | 0.19 (0.10) | 0.35 (0.22)
  Extension Month 21 (n=154, 166) | 0.19 (0.11) | 0.35 (0.22)
  Extension Month 24 (n=150, 156) | 0.20 (0.11) | 0.36 (0.24)
  Extension Month 27 (n=142, 153) | 0.20 (0.11) | 0.36 (0.23)
  Extension Month 30 (n=141, 149) | 0.20 (0.11) | 0.37 (0.24)
  Extension Month 33 (n=133, 144) | 0.20 (0.12) | 0.36 (0.24)
  Extension Month 36 (n=113, 136) | 0.21 (0.11) | 0.36 (0.25)
  Extension Month 39 (n=57, 67) | 0.23 (0.14) | 0.39 (0.23)

12. Secondary Outcome: Baseline Dyspnea Index (BDI)
Description: Clinician administered instrument to measure the baseline severity of breathlessness (shortness of breath) in symptomatic patients with 3 domains: functional impairment, magnitude of task, and magnitude of effort. BDI score range 0 (very severe impairment) to 4 (no impairment) scaled to a BDI focal score (0-12). Lower score indicates greater impairment.
Time Frame: Week - 1
Population: FAS FEV1. Due to early termination of the study a limited set of analyses were undertaken and results of the Baseline Dyspnea Index were not summarized as planned.
Measure: Mean (Standard Deviation); unit: scores on scale
Arm/Group | Inhaled Insulin | Subcutaneous Insulin
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Transition Dyspnea Index (TDI)
Description: Clinician administered instrument to measure the baseline severity of breathlessness (shortness of breath) in symptomatic patients with 3 domains: functional impairment, magnitude of task, and magnitude of effort. TDI score range -3 (major deterioration) to +3 (major improvement); sum of all domains yields the TDI focal score (-9 to +9); lower score indicates greater deterioration. Compared to previous scoring to determine deterioration or improvement.
Time Frame: Week 4 through ,Extension Follow-up Month 6 and every 6 months thereafter or end of study
Population: FAS FEV1. Due to early termination of the study a limited set of analyses were undertaken and results of the Transition Dyspnea Index were not summarized as planned.
Measure: Mean (Standard Deviation); unit: scores on scale
Arm/Group | Inhaled Insulin | Subcutaneous Insulin
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Lipids
Description: Total cholesterol, high-density lipoprotein (HDL) cholesterol, low-density lipoprotein (LDL) cholesterol, and triglycerides measured as milligrams per deciliter (mg/dL).
Time Frame: Week -4 through Month 24
Population: Full Analysis Set (FAS): received at least 1 dose of study treatment. Due to early termination of the study a limited set of analyses were undertaken and lipid results were not summarized as planned.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Inhaled Insulin | Subcutaneous Insulin
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Cough Questionnaire
Description: Subject completed cough questionnaire with reference to the past 4 weeks. Six question instrument to measure cough frequency (night, day), severity, timing in relation to short-acting insulin dosing, severity related to insulin dosing (subcutaneous [SC] or inhaled), and productivity of cough; range 0 (no symptoms) to 4 (severe symptoms). Questionnaire was administered at Week 0 and then at subsequent visits only if cough was identified as an adverse event not explained by a concomitant condition, such as an upper respiratory tract infection.
Time Frame: Week 0 and if indicated through Extension Follow up Month 3
Population: FAS. Due to early termination of the study a limited set of analyses were undertaken and results of the Cough Questionnaire were not summarized as planned.
Measure: Mean (Standard Deviation); unit: scores on scale
Arm/Group | Inhaled Insulin | Subcutaneous Insulin
Number analyzed (Participants) | 0 | 0

16. Primary Outcome: Change From Baseline in Carbon Monoxide Diffusion Capacity (DLco)
Description: Change from Baseline: mean of (value of Carbon Monoxide Diffusing Capacity [DLco] measured in milliters/minutes/millimeters of mercury [mL/min/mmHg] at observation minus Baseline value).
Time Frame: Baseline through Extension Follow-up Month 3
Population: FAS FEV1; (n) = number of subjects with analyzable data at observation for inhaled insulin and SC insulin, respectively. Due to study termination, originally planned inferential analysis change from Month 3 to extension Month 60 was not done.
Measure: Mean (Standard Deviation); unit: mL/min/mmHg
Arm/Group | Inhaled Insulin | Subcutaneous Insulin
Number analyzed (Participants) | 283 | 281
mL/min/mmHg
  Baseline (n=283, 281) | 28.09 (6.20) | 27.18 (6.40)
  Month 3 (n=277, 264) | -1.09 (1.73) | -0.29 (1.71)
  Month 6 (n=262, 273) | -1.17 (2.16) | -0.26 (1.85)
  Month 9 (n=250, 266) | -1.16 (2.09) | -0.41 (1.91)
  Month 12 (n=241, 258) | -1.40 (2.15) | -0.41 (2.15)
  Month 15 (n=235, 249) | -1.16 (2.17) | -0.42 (2.17)
  Month 18 (n=227, 232) | -1.21 (2.28) | -0.45 (2.22)
  Month 21 (n=218, 224) | -1.29 (2.49) | -0.56 (2.07)
  Month 24 (n=208, 219) | -1.28 (2.29) | -0.71 (2.40)
  Follow-up Month 1 (n=242,208) | -0.81 (2.20) | -0.81 (2.42)
  Follow-up Month 3 (n=247,225) | -0.77 (2.46) | -0.80 (2.10)
  Follow-up Month 6 (n=240,218) | -0.77 (2.36) | -0.67 (2.28)
  Extension Month 1 (n=166,175) | -1.15 (2.54) | -0.55 (2.35)
  Extension Month 3 (n=161,173) | -1.43 (2.37) | -0.73 (2.45)
  Extension Month 6 (n=158,169) | -1.38 (2.37) | -0.78 (2.54)
  Extension Month 9 (n=151,163) | -1.17 (2.52) | -0.74 (2.57)
  Extension Month 12 (n=152,161) | -1.70 (2.46) | -0.70 (2.60)
  Extension Month 15 (n=143,160) | -1.70 (2.27) | -0.72 (2.94)
  Extension Month 18 (n=148,159) | -1.67 (2.36) | -1.02 (2.72)
  Extension Month 21 (n=144,156) | -1.51 (2.59) | -0.88 (2.64)
  Extension Month 24 (n=140,152) | -1.63 (2.46) | -0.70 (2.72)
  Extension Month 27 (n=136,144) | -1.25 (2.65) | -0.76 (2.75)
  Extension Month 30 (n=135,146) | -1.36 (2.54) | -0.75 (2.59)
  Extension Month 33 (n=127,139) | -1.31 (2.54) | -0.81 (2.55)
  Extension Month 36 (n=105,122) | -1.53 (2.53) | -0.96 (2.82)
  Extension Month 39 (n=52, 64) | -2.02 (3.72) | -0.93 (2.59)
  Extension Month 39 (LOCF) (n=177, 187) | -1.66 (2.90) | -0.90 (2.55)
  Extension Follow Up Month 3 (n=115, 101) | -0.89 (2.35) | -1.11 (2.59)
Statistical Analysis 1: Comparison: Inhaled Insulin vs Subcutaneous Insulin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.744, 90% CI [-0.981 to -0.506], Standard Error of Mean 0.144
Statistical Analysis 2: Comparison: Inhaled Insulin vs Subcutaneous Insulin; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.797, 90% CI [-1.073 to -0.522], Standard Error of Mean 0.167
Statistical Analysis 3: Comparison: Inhaled Insulin vs Subcutaneous Insulin; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.667, 90% CI [-0.949 to -0.384], Standard Error of Mean 0.171
Statistical Analysis 4: Comparison: Inhaled Insulin vs Subcutaneous Insulin; [analysis description as in outcome 1, analysis 4]; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.826, 90% CI [-1.123 to -0.528], Standard Error of Mean 0.181
Statistical Analysis 5: Comparison: Inhaled Insulin vs Subcutaneous Insulin; [analysis description as in outcome 1, analysis 5]; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.610, 90% CI [-0.923 to -0.296], Standard Error of Mean 0.190
Statistical Analysis 6: Comparison: Inhaled Insulin vs Subcutaneous Insulin; [analysis description as in outcome 1, analysis 6]; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.577, 90% CI [-0.910 to -0.245], Standard Error of Mean 0.202
Statistical Analysis 7: Comparison: Inhaled Insulin vs Subcutaneous Insulin; [analysis description as in outcome 1, analysis 7]; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.613, 90% CI [-0.962 to -0.263], Standard Error of Mean 0.212
Statistical Analysis 8: Comparison: Inhaled Insulin vs Subcutaneous Insulin; [analysis description as in outcome 1, analysis 8]; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.385, 90% CI [-0.736 to -0.034], Standard Error of Mean 0.213
Statistical Analysis 9: Comparison: Inhaled Insulin vs Subcutaneous Insulin; [analysis description as in outcome 1, analysis 9]; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.150, 90% CI [-0.197 to 0.497], Standard Error of Mean 0.211
Statistical Analysis 10: Comparison: Inhaled Insulin vs Subcutaneous Insulin; [analysis description as in outcome 1, analysis 10]; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.166, 90% CI [-0.160 to 0.492], Standard Error of Mean 0.198
Statistical Analysis 11: Comparison: Inhaled Insulin vs Subcutaneous Insulin; [analysis description as in outcome 1, analysis 11]; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = 0.069, 90% CI [-0.274 to 0.411], Standard Error of Mean 0.208
Statistical Analysis 12: Comparison: Inhaled Insulin vs Subcutaneous Insulin; [analysis description as in outcome 1, analysis 12]; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.460, 90% CI [-0.876 to -0.043], Standard Error of Mean 0.252
Statistical Analysis 13: Comparison: Inhaled Insulin vs Subcutaneous Insulin; [analysis description as in outcome 1, analysis 13]; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.579, 90% CI [-0.986 to -0.172], Standard Error of Mean 0.247
Statistical Analysis 14: Comparison: Inhaled Insulin vs Subcutaneous Insulin; [analysis description as in outcome 1, analysis 14]; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.460, 90% CI [-0.880 to -0.040], Standard Error of Mean 0.255
Statistical Analysis 15: Comparison: Inhaled Insulin vs Subcutaneous Insulin; [analysis description as in outcome 1, analysis 15]; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.385, 90% CI [-0.822 to 0.053], Standard Error of Mean 0.265
Statistical Analysis 16: Comparison: Inhaled Insulin vs Subcutaneous Insulin; [analysis description as in outcome 1, analysis 16]; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.930, 90% CI [-1.372 to -0.487], Standard Error of Mean 0.268
Statistical Analysis 17: Comparison: Inhaled Insulin vs Subcutaneous Insulin; [analysis description as in outcome 1, analysis 17]; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.823, 90% CI [-1.296 to -0.351], Standard Error of Mean 0.286
Statistical Analysis 18: Comparison: Inhaled Insulin vs Subcutaneous Insulin; [analysis description as in outcome 1, analysis 18]; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.525, 90% CI [-0.965 to -0.084], Standard Error of Mean 0.267
Statistical Analysis 19: Comparison: Inhaled Insulin vs Subcutaneous Insulin; [analysis description as in outcome 1, analysis 19]; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.647, 90% CI [-1.104 to -0.191], Standard Error of Mean 0.276
Statistical Analysis 20: Comparison: Inhaled Insulin vs Subcutaneous Insulin; [analysis description as in outcome 1, analysis 20]; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.853, 90% CI [-1.340 to -0.367], Standard Error of Mean 0.295
Statistical Analysis 21: Comparison: Inhaled Insulin vs Subcutaneous Insulin; [analysis description as in outcome 1, analysis 21]; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.390, 90% CI [-0.890 to 0.111], Standard Error of Mean 0.303
Statistical Analysis 22: Comparison: Inhaled Insulin vs Subcutaneous Insulin; [analysis description as in outcome 1, analysis 22]; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.636, 90% CI [-1.119 to -0.153], Standard Error of Mean 0.293
Statistical Analysis 23: Comparison: Inhaled Insulin vs Subcutaneous Insulin; [analysis description as in outcome 1, analysis 23]; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.522, 90% CI [-1.000 to -0.043], Standard Error of Mean 0.290
Statistical Analysis 24: Comparison: Inhaled Insulin vs Subcutaneous Insulin; [analysis description as in outcome 1, analysis 24]; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.744, 90% CI [-1.315 to -0.173], Standard Error of Mean 0.346
Statistical Analysis 25: Comparison: Inhaled Insulin vs Subcutaneous Insulin; [analysis description as in outcome 1, analysis 25]; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -1.378, 90% CI [-2.420 to -0.335], Standard Error of Mean 0.628
Statistical Analysis 26: Comparison: Inhaled Insulin vs Subcutaneous Insulin; [analysis description as in outcome 1, analysis 26]; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.720, 90% CI [-1.183 to -0.258], Standard Error of Mean 0.280
Statistical Analysis 27: Comparison: Inhaled Insulin vs Subcutaneous Insulin; [analysis description as in outcome 1, analysis 27]; Test type: Superiority or Other; ANCOVA; Mean Difference (Final Values) = -0.061, 90% CI [-0.594 to 0.472], Standard Error of Mean 0.323

17. Primary Outcome: Summary of ≥ 20% Decliners in Carbon Monoxide Diffusing Capacity (DLco).
Description: Number of subjects with a post-baseline Carbon Monoxide Diffusing Capacity (DLco) decrease of ≥ 20% [(baseline observed value minus visit observed value)/(baseline observed value) * 100]; in the absence of an obvious intercurrent illness, a repeat DLco was performed.
Time Frame: Month 3 through Extension Follow-up Month 3
Population: FAS FEV1; (n) = number of subjects with analyzable data at observation for inhaled insulin and SC insulin, respectively.
Measure: Number; unit: participants
Arm/Group | Inhaled Insulin | Subcutaneous Insulin
Number analyzed (Participants) | 283 | 281
participants
  Month 3 (n=277, 264) | 0 | 1
  Month 6 (n=262, 273) | 1 | 0
  Month 9 (n=250, 266) | 2 | 1
  Month 12 (n=241, 258) | 2 | 1
  Month 15 (n=235, 249) | 1 | 2
  Month 18 (n=227, 232) | 5 | 4
  Month 21 (n=218, 224) | 4 | 2
  Month 24 (n=208, 219) | 2 | 2
  Follow-up Month 1 (n=242, 208) | 3 | 3
  Follow-up Month 3 (n=247, 225) | 1 | 1
  Follow-up Month 6 (n=240, 218) | 1 | 2
  Extension Month 1 (n=166, 175) | 5 | 0
  Extension Month 3 (n=161, 173) | 4 | 1
  Extension Month 6 (n=158, 169) | 4 | 2
  Extension Month 9 (n=151, 163) | 2 | 2
  Extension Month 12 (n=152, 161) | 5 | 2
  Extension Month 15 (n=143, 160) | 3 | 2
  Extension Month 18 (n=148, 159) | 1 | 4
  Extension Month 21 (n=144, 156) | 5 | 3
  Extension Month 24 (n=140, 152) | 5 | 1
  Extension Month 27 (n=136, 144) | 4 | 2
  Extension Month 30 (n=135, 146) | 4 | 4
  Extension Month 33 (n=127, 139) | 3 | 2
  Extension Month 36 (n=105, 122) | 4 | 7
  Extension Month 39 (n=52, 64) | 3 | 1
  Extension Follow Up Month 3 (n=115, 101) | 3 | 2

18. Secondary Outcome: Forced Vital Capacity (FVC)
Description: Forced Vital Capacity (FVC) measured in liters (L).
Time Frame: Week -3 through Extension Follow-up Month 6 or End of Study
Population: FAS FEV1. Due to early termination of the study a limited set of analyses were undertaken and FVC results were not summarized as planned.
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Inhaled Insulin | Subcutaneous Insulin
Number analyzed (Participants) | 0 | 0

19. Secondary Outcome: Total Lung Capacity (TLC)
Description: Total Lung Capacity measured in liters (L).
Time Frame: Week -3 through Extension Follow-up Month 6 or End of Study
Population: FAS FEV1. Due to early termination of the study a limited set of analyses were undertaken and TLC results were not summarized as planned.
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Inhaled Insulin | Subcutaneous Insulin
Number analyzed (Participants) | 0 | 0

20. Primary Outcome: Annual Rate of Change in Forced Expiratory Volume in 1 Second (FEV1)
Description: Annual rate of change in FEV1 calculated as slope over time [visit] for forced expiratory volume in 1 second measured as liters per year (L/yr).
Time Frame: Week -2 through Extension Follow-up Month 6 or end of study
Population: FAS FEV1. Due to early termination of the study a limited set of analyses were undertaken and results of the Annual Rate of Change in FEV1 were not summarized as planned.
Measure: Mean (Standard Deviation); unit: liters per year
Arm/Group | Inhaled Insulin | Subcutaneous Insulin
Number analyzed (Participants) | 0 | 0

21. Primary Outcome: Annual Rate of Change in Carbon Monoxide Diffusion Capacity (DLco)
Description: Annual rate of change in DLco calculated as slope over time (visit) measured as milliliters per minute per millimeters of hemoglobin per year (ml/min/mmHg/yr).
Time Frame: Week -2 through Extension Follow-up Month 6 or end of study
Population: FAS FEV1. Due to early termination of the study a limited set of analyses were undertaken and results of the annual rate of change in DLco were not summarized as planned.
Measure: Mean (Standard Deviation); unit: ml/min/mmHg/yr
Arm/Group | Inhaled Insulin | Subcutaneous Insulin
Number analyzed (Participants) | 0 | 0

22. Secondary Outcome: Insulin Antibodies
Description: Median insulin antibodies at each visit measured in micro units per milliliter (microU/mL).
Time Frame: Baseline through Extension Month 39
Population: FAS; (n)= number of subjects with analyzable data at observation: inhaled insulin/SC insulin, respectively. Insulin antibody levels increased in Exubera®-treated compared to control subjects; results are included to establish there were no safety consequences due to these elevations although this was not an originally specified protocol endpoint.
Measure: Median (Full Range); unit: microU/mL
Arm/Group | Inhaled Insulin | Subcutaneous Insulin
Number analyzed (Participants) | 284 | 283
microU/mL
  Baseline (n=284, 283) | 4.50 [1.05 to 3514.00] | 4.10 [1.05 to 1324.00]
  Week 3 (n=262, 260) | 7.50 [1.05 to 6056.00] | 3.60 [1.05 to 828.00]
  Week 6 (n=267, 260) | 15.00 [1.05 to 12445.00] | 4.00 [1.05 to 1792.00]
  Month 3 (n=271, 274) | 31.00 [1.05 to 4108.00] | 4.25 [1.05 to 876.00]
  Week 18 (n=263, 271) | 49.00 [1.05 to 1968.00] | 4.40 [1.05 to 1012.00]
  Month 6 (n=254, 268) | 88.50 [1.05 to 1420.00] | 5.10 [1.05 to 1352.00]
  Month 9 (n=244, 262) | 134.50 [1.05 to 2776.00] | 4.95 [1.05 to 1608.00]
  Month 12 (n=234, 258) | 142.50 [1.05 to 3156.00] | 4.90 [1.05 to 2192.00]
  Month 15 (n=230, 250) | 109.50 [1.05 to 4380.00] | 4.70 [1.05 to 1360.00]
  Month 18 (n=226, 233) | 91.00 [1.05 to 2390.00] | 4.40 [1.05 to 1655.00]
  Month 21 (n=216, 228) | 59.50 [1.05 to 2575.00] | 3.85 [1.05 to 932.00]
  Month 24 (n=212, 224) | 67.00 [1.05 to 2360.00] | 4.40 [1.05 to 1420.00]
  Follow-up Month 1 (n=234, 209) | 41.50 [1.05 to 27286.00] | 4.20 [1.05 to 1285.00]
  Follow-up Month 3 (n=245, 226) | 28.00 [1.05 to 8119.00] | 4.20 [1.05 to 382.00]
  Follow-up Month 6 (n=239, 223) | 22.00 [1.05 to 5280.00] | 4.40 [1.05 to 1265.00]
  Extension Month 1 (n=164, 176) | 37.50 [1.05 to 3985.00] | 4.50 [1.05 to 900.00]
  Extension Month 3 (165, 177) | 45.00 [1.05 to 3405.00] | 4.40 [1.05 to 1260.00]
  Extension Month 6 (n=162, 176) | 42.50 [1.05 to 3145.00] | 3.55 [1.05 to 720.00]
  Extension Month 9 (n=154, 167) | 41.00 [1.05 to 2465.00] | 4.70 [1.05 to 873.00]
  Extension Month 12 (n=155, 167) | 49.00 [1.05 to 3280.00] | 4.30 [1.05 to 1310.00]
  Extension Month 15 (n=149, 163) | 43.00 [1.05 to 3955.00] | 4.50 [1.05 to 1330.00]
  Extension Month 18 (n=149, 160) | 45.00 [1.05 to 10755.00] | 3.60 [1.05 to 1430.00]
  Extension Month 21 (n=151, 157) | 44.00 [1.05 to 3200.00] | 3.60 [1.05 to 820.00]
  Extension Month 24 (n=146, 153) | 42.50 [1.05 to 3920.00] | 4.40 [1.05 to 758.00]
  Extension Month 27 (n=138, 148) | 35.00 [1.05 to 3040.00] | 6.35 [1.05 to 1121.00]
  Extension Month 30 (n=139, 150) | 36.00 [1.05 to 3730.00] | 5.25 [1.05 to 1110.00]
  Extension Month 33 (n=129, 142) | 35.00 [1.05 to 3980.00] | 4.30 [1.05 to 845.00]
  Extension Month 36 (n=104, 132) | 30.50 [1.05 to 1477.00] | 3.65 [1.05 to 876.00]
  Extension Month 39 (n=54, 66) | 25.50 [1.05 to 1750.00] | 1.58 [1.05 to 742.00]

ADVERSE EVENTS:
Description: Adverse events for this study are reported using MedDRA in these Basic Results, but are reported using COSTART in the Clinical Study Report and PhRMA Web Synopsis for consistency with earlier studies. Consequently, subtle differences may be observed.
Arm/Group | Inhaled Insulin | Subcutaneous Insulin
Serious Adverse Events (participants affected / at risk) | 50/290 | 65/290
Other Adverse Events (participants affected / at risk) | 290/290 | 289/290
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Inhaled Insulin (N=290) | Subcutaneous Insulin (N=290)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 4
Coronary artery stenosis (Cardiac disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Macular degeneration (Eye disorders) | 1 | 0
Retinal detachment (Eye disorders) | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Colonic polyp (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Peptic ulcer (Gastrointestinal disorders) | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 1 | 0
Chest discomfort (General disorders) | 1 | 0
Chest pain (General disorders) | 4 | 2
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 2 | 1
Appendicitis (Infections and infestations) | 0 | 2
Cellulitis (Infections and infestations) | 1 | 1
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 1 | 0
Gangrene (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 1
Histoplasmosis (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Kidney infection (Infections and infestations) | 1 | 0
Meningitis (Infections and infestations) | 0 | 1
Necrotising fasciitis (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 2
Postoperative wound infection (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 2 | 0
Bone fissure (Injury, poisoning and procedural complications) | 0 | 1
Burns first degree (Injury, poisoning and procedural complications) | 0 | 1
Burns second degree (Injury, poisoning and procedural complications) | 0 | 1
Burns third degree (Injury, poisoning and procedural complications) | 1 | 1
Face injury (Injury, poisoning and procedural complications) | 0 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 1
Jaw fracture (Injury, poisoning and procedural complications) | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Diabetic foot (Metabolism and nutrition disorders) | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 17 | 26
Ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 0 | 1
Grand mal convulsion (Nervous system disorders) | 0 | 1
Intracranial hypotension (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 2
Sciatica (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 2
Major depression (Psychiatric disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 1
Renal colic (Renal and urinary disorders) | 1 | 1
Ureteric obstruction (Renal and urinary disorders) | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 1 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1
Uterine disorder (Reproductive system and breast disorders) | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Ileostomy (Surgical and medical procedures) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Inhaled Insulin (N=290) | Subcutaneous Insulin (N=290)
Abdominal pain upper (Gastrointestinal disorders) | 10 | 17
Diarrhoea (Gastrointestinal disorders) | 36 | 28
Nausea (Gastrointestinal disorders) | 30 | 21
Vomiting (Gastrointestinal disorders) | 20 | 17
Asthenia (General disorders) | 19 | 21
Chest pain (General disorders) | 18 | 17
Fatigue (General disorders) | 22 | 25
Seasonal allergy (Immune system disorders) | 15 | 15
Bronchitis (Infections and infestations) | 24 | 25
Gastroenteritis (Infections and infestations) | 29 | 25
Gastroenteritis viral (Infections and infestations) | 26 | 18
Influenza (Infections and infestations) | 84 | 85
Nasopharyngitis (Infections and infestations) | 96 | 111
Pharyngitis (Infections and infestations) | 15 | 17
Rhinitis (Infections and infestations) | 20 | 14
Sinusitis (Infections and infestations) | 50 | 47
Upper respiratory tract infection (Infections and infestations) | 124 | 105
Urinary tract infection (Infections and infestations) | 31 | 32
Contusion (Injury, poisoning and procedural complications) | 7 | 15
Hyperlipidaemia (Metabolism and nutrition disorders) | 17 | 7
Hypoglycaemia (Metabolism and nutrition disorders) | 282 | 285
Arthralgia (Musculoskeletal and connective tissue disorders) | 31 | 34
Back pain (Musculoskeletal and connective tissue disorders) | 24 | 31
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 17 | 24
Pain in extremity (Musculoskeletal and connective tissue disorders) | 18 | 30
Tendonitis (Musculoskeletal and connective tissue disorders) | 16 | 13
Dizziness (Nervous system disorders) | 20 | 22
Headache (Nervous system disorders) | 41 | 46
Tremor (Nervous system disorders) | 42 | 43
Depression (Psychiatric disorders) | 12 | 25
Insomnia (Psychiatric disorders) | 16 | 8
Stress (Psychiatric disorders) | 17 | 15
Cough (Respiratory, thoracic and mediastinal disorders) | 130 | 53
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 24 | 6
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 21 | 14
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 35 | 47
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 12 | 15
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 25 | 23
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 28 | 31
Hypertension (Vascular disorders) | 24 | 24

LIMITATIONS AND CAVEATS:
Due to early termination of study, none of the subjects completed the study as planned. Subjects active at the time of study termination completed an end-of-study assessment and a 3-month follow-up visit.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.